CLINICAL TRIAL: NCT05980715
Title: A Randomized Controlled, Non-inferior, Phase III Study of PD-1 Inhibitor Therapy Versus Radiotherapy in pCR Patients With Locally Advanced Head and Neck Squamous Cell Carcinoma After Neoadjuvant Immunochemotherapy
Brief Title: PD-1 Inhibitor Therapy Versus Radiotherapy in pCR Patients With Locally Advanced HNSCC After Neoadjuvant Immunochemotherapy
Acronym: HNC-SYSU-003
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First People's Hospital of Foshan (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Affiliated Cancer Hospital of Shantou University Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2023-463-02
Record Dates: First submitted 2023-06-05; First posted 2023-08-08 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: HNSCC; Radiotherapy; PD-1
Keywords: HNSCC; radiotherapy; PD-1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1（PD-1） (Experimental): Radiotherapy free treatment: the experimental group took PD-1 inhibitor maintenance regimen.
  Interventions: Drug: PD-1inhibitor
- Arm 2（radiotherapy） (Active Comparator): conventional radiotherapy (chemoradiotherapy) regimen, and received comprehensive treatment according to the guidelines (radiotherapy or platinum-based concurrent chemoradiotherapy as stipulated in the guidelines).
  Interventions: Radiation: concurrent chemoradiotherapy

INTERVENTIONS:
Drug: PD-1inhibitor — The PD-1 monoclonal antibody was the same as the neoadjuvant therapy before surgery, and the postoperative level was maintained at Q3*6.
  Arms: Arm 1（PD-1）
Radiation: concurrent chemoradiotherapy — According to the guidelines, concurrent chemoradiotherapy is required, and carboplatin (50mg/m2) plus concurrent radiotherapy or cisplatin (30mg/m2) plus concurrent radiotherapy is optional.
  Arms: Arm 2（radiotherapy）

SUMMARY:
In patients with locally advanced head and neck squamous cell carcinoma undergoing standard surgical treatment after neoadjuvant immunochemotherapy, can PD-1 inhibitor therapy be used instead of adjuvant radiotherapy for both primary and lymph node pathology? To provide further evidence-based medical evidence for the late precision treatment of HNSCC patients after neoadjuvant immunochemotherapy. Avoid the side effects caused by excessive radiotherapy, especially avoid the occurrence of second primary cancer, radiation osteonecrosis and other diseases.

1. Main study endpoint:

   A randomized controlled, non-inferiority, multicentre Phase III trial was conducted to investigate the difference in 5-year overall survival (OS) between experimental group (Group B) and control group (group A) in patients undergoing standard surgical treatment after neoadjuvant immunochemotherapy for locally advanced HNSCC, with both primary and lymph node pathology revealed by pCR. At the same time, adverse events and safety were evaluated according to NCI-CTCAE 5.0 criteria and RTOG later radiotherapy damage evaluation criteria.

   Safety indicators focused on late radiotherapy toxicity and the incidence of grade 3 and 4 adverse reactions in NCI-CTC AE 5.0 and RTOG. The differences in the incidence of grade 3 and 4 adverse events were compared between the experimental group and the control group.
2. Secondary study endpoint:

The differences in 2-year disease-free survival (DFS), regional relapse-free survival (RRFS), distant metastasis free survival (DMFS), safety and adverse events were compared.

Safety evaluation NCI-CTC AE 5.0 standard was used to evaluate the acute safety index of radiotherapy, and RTOG late-stage damage evaluation standard was used to evaluate the late-stage safety index of radiotherapy.

4) Exploratory goals The influence of prognostic laboratory indicators, clinical risk factors were analyzed. To explore the factors that influence the efficacy of radiotherapy after pCR immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* In this study, patients with locally advanced head and neck squamous cell carcinoma (AJCC 8th) who underwent standard surgical treatment after neoadjuvant immunochemotherapy and showed pCR in both primary lesions and lymph node pathology were selected. Locally advanced squamous cell carcinoma of head and neck includes: i) T3, N0, M0; 2) T1-T3, N1-N2, M0; 3) T4a, N0-2, M0.
* No history of other malignant tumors
* Ages 18-65
* Normal baseline inspection:

  1. The absolute value of neutrophil granulocyte (ANC) ≥1.5x109/L in the last 14 days without the use of granulocyte colony stimulating factor;
  2. Platelets ≥100×109/L without blood transfusion in the past 14 days;
  3. Hemoglobin &gt without blood transfusion or use of erythropoietin within the last 14 days; 9g/dL;
  4. Total bilirubin ≤1.5× upper limit of normal value (ULN);
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (ALT or AST ≤5×ULN in patients with liver metastasis);
  6. Serum creatinine ≤1.5×ULN and creatinine clearance (calculated by Cockcroft-Gault formula) ≥60 ml/min;
  7. Good coagulation function, defined as International Standardized ratio (INR) or prothrombin time (PT) ≤1.5 times ULN;
  8. Normal thyroid function, defined as thyroid stimulating hormone (TSH) within the normal range. Subjects whose baseline TSH is outside the normal range can be enrolled if total T3 (or FT3) and FT4 are within the normal range;
  9. The myocardial enzyme profile was within the normal range (if the researchers comprehensively judged that the simple laboratory abnormality was not clinically significant, it was also allowed to be included);
  10. For female subjects of childbearing age, a urine or serum pregnancy test should be tested negative within 3 days prior to receiving the first study drug administration (day 1 of Cycle 1). If the urine pregnancy test results cannot be confirmed negative, a blood pregnancy test is requested. Women of non-reproductive age were defined as at least one year after menopause or having undergone surgical sterilization or hysterectomy;
  11. If there is a risk of conception, all subjects (male or female) shall use contraception with an annual failure rate of less than 1% for the entire duration of treatment up to 120 days after the last study drug administration (or 180 days after the last chemotherapeutic drug administration).

  5 Sign informed consent

Exclusion Criteria:

* 1 HNSCC is not the initial diagnosis of other malignant tumors or neoadjuvant therapy.
* Prior to treatment An active autoimmune immune disease requiring systemic therapy (e.g. the use of disease-modifying drugs, glucocorticoids, or immunosuppressants) has occurred in the last 2 years. Alternative therapies (such as thyroxine, insulin, or physiologic glucocorticoids for adrenal or pituitary insufficiency) are not considered systemic therapy;
* Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
* Known history of human immunodeficiency virus (HIV) infection (i.e. HIV 1/2 antibody positive);
* Untreated active hepatitis B (defined as HBsAg positive and HBV-DNA copy number detected greater than the upper limit of normal value in the laboratory of the study center);

Note: Hepatitis B subjects who meet the following criteria can also be enrolled:

1) HBV viral load &lt before initial administration; At 1000 copies /ml (200 IU/ml), subjects should receive anti-HBV therapy to avoid viral reactivation throughout the study treatment period 2) For subjects with anti-HBC (+), HBsAg (-), anti-HBS (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring of viral reactivation is required

* Active HCV infected subjects (HCV antibody positive and HCV-RNA level above the lower limit);
* Pregnant or lactating women;
* The presence of any serious or uncontrolled systemic disease, such as:

  1. The resting electrocardiogram (ECG) presents significant and severely uncontrollable abnormalities in rhythm, conduction or morphology, such as complete left bundle branch block, Ⅱ degree or above heart block, ventricular arrhythmia or atrial fibrillation;
  2. Unstable angina pectoris, congestive heart failure, and NYHA grade ≥ 2 chronic heart failure;
  3. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, occurred within 6 months before treatment;
  4. Poor blood pressure control (systolic > 140 mmHg, diastolic > 90 mmHg);
  5. A history of non-infectious pneumonia requiring glucocorticoid therapy or clinically active interstitial lung disease within 1 year prior to initial administration;
  6. Active pulmonary tuberculosis;
  7. There is an active or uncontrolled infection that requires systemic treatment;
  8. Clinically active diverticulitis, abdominal abscess, gastrointestinal obstruction;
  9. Liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
  10. Poor diabetes control (fasting blood glucose (FBG) > 10mmol/L);
  11. Urine routine indicated urine protein ≥++, and confirmed 24 hours urine protein quantity > 1.0 g;
  12. Patients with mental disorders and unable to cooperate with treatment;
* Medical history or evidence of disease that may interfere with test results, prevent subjects from fully participating in the study, abnormal values of treatment or laboratory tests, or other conditions that the investigator considers unsuitable for enrollment. The investigator considers other potential risks unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) | 5 years
  Overall survival(OS) is the time from day 1 of study treatment(the time randomized) until death from any cause.
The percentage of Grade 3 and 4 adverse reactions in NCI-CTC AE 5.0 and RTOG | 5 years
  The incidence(percentage) of late toxicity , Grade 3 and 4 adverse reactions in NCI-CTC AE 5.0 and RTOG.

SECONDARY OUTCOMES:
Disease-free survival （DFS） | 2 years
  DFS(by months) is defined as the time from treatment until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from treatment or receives another anti-cancer therapy prior to disease DFS is defined as the time from treatment until the date of the first relapse (local/regional recurrence or distant metastasis) or death (from any cause) whichever comes firsts and regardless of whether the patient withdraws from treatment or receives another anti-cancer therapy prior to disease relapse.
regional recurrence-free survival (RRFS) | 2 years
  The time( by months) from randomization to clinically confirmed recurrence in the lymph node drainage area. Deaths were counted in RRFS.
distant metastasis free survival (DMFS) | 2 years
  The time( by months) from randomization to clinically confirmed distant metastasis.
Number and percentage of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v5.0 and RTOG | 2 years
  The detail number and percentage of adverse events by every systems Assessed by CTCAE v5.0 and RTOG.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun yat-sen memorial hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No